CLINICAL TRIAL: NCT00270920
Title: A Randomised Controlled Trial to Compare Antenatal Preparation and Postnatal Counseling Strategies for Improving Breastfeeding Rates
Brief Title: A Randomised Controlled Trial to Compare Antenatal Preparation and Postnatal Counseling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: NUS IRB 03003; NHG RPR 03002
Record Dates: First submitted 2005-12-28; First posted 2005-12-29 (Estimated); Last update posted 2008-07-15 (Estimated); Status verified 2008-07

CONDITIONS: Breastfeeding
Keywords: Initiation, Maintenance, Breastfeeding
MeSH Terms: conditions — Breast Feeding

INTERVENTIONS:
Behavioral: Lactation counseling

SUMMARY:
This is a randomised controlled trial to compare antenatal preparation and postnatal counseling strategies for improving breastfeeding rates.

The objectives are:

1. to study the effect of a standard two-encounter postnatal lactation counseling protocol on the initiation and maintenance of exclusive breastfeediing in mothers
2. to compare the effect of a standard two-encounter postnatal lactation counseling protocol with a single-encounter antenatal breastfeeding education protocol on the initiation and maintenance of exclusive breastfeeding in mothers.

DETAILED DESCRIPTION:
All pregnant mothers who wish to breastfeed after 34 weeks of gestation, and who do not have a high risk pregnancy as determined by investigator or have a multiple pregnancy in current pregnancy and have given their written informed consent will be randomised into three groups. Group 1 will receive standard hospital care. Group 2 will receive 1 session of antenatal counseling and Group 3 will receive 2 sessions of postanatal lactation counseling. All will receive postnatal follow up phone calls using questions from Case Report Forms at 2 weeks, 8 weeks, 3 months, 6 months and 12 months. The mothers who are not contactable for 3 consecutive months will be withdrawn from the study.

ELIGIBILITY:
Inclusion Criteria:

Pregnant woman who wants to breastfeed her child after 34 weeks of gestation and written informed consent given

Exclusion Criteria:

Pregnant women with high risk pregnancy as determined by the investigator.

-

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 450
Dates: Start 2004-02; Study Completion 2006-03

PRIMARY OUTCOMES:
Study the effect of a standard two-encounter postnatal lactation counseling protocol on the initiation and maintenance of exclusive breastfeeding in mothers

SECONDARY OUTCOMES:
Compare the effect of a standard two-encounter postnatal lactation counseling protocol with a single-encounter antenatal breastfeeding education protocol on the initiation and maintenance of exclusive breastfeeding in mothers.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Rauff, MBBS, FRCOG, Principal Investigator — National University of Singapore /National University Hospital
Locations (1):
- National University Hospital, Singapore, Singapore

REFERENCES:
- [Background] Morrow AL, Guerrero ML, Shults J, Calva JJ, Lutter C, Bravo J, Ruiz-Palacios G, Morrow RC, Butterfoss FD. Efficacy of home-based peer counselling to promote exclusive breastfeeding: a randomised controlled trial. Lancet. 1999 Apr 10;353(9160):1226-31. doi: 10.1016/S0140-6736(98)08037-4. PMID 10217083
- [Result] Haider R, Ashworth A, Kabir I, Huttly SR. Effect of community-based peer counsellors on exclusive breastfeeding practices in Dhaka, Bangladesh: a randomised controlled trial [see commments]. Lancet. 2000 Nov 11;356(9242):1643-7. doi: 10.1016/s0140-6736(00)03159-7. PMID 11089824
- [Derived] Su LL, Chong YS, Chan YH, Chan YS, Fok D, Tun KT, Ng FS, Rauff M. Antenatal education and postnatal support strategies for improving rates of exclusive breast feeding: randomised controlled trial. BMJ. 2007 Sep 22;335(7620):596. doi: 10.1136/bmj.39279.656343.55. Epub 2007 Aug 1. PMID 17670909